CLINICAL TRIAL: NCT00353834
Title: The Effect of Exenatide Compared to Lantus Insulin on Vascular Function Before and After a Meal Tolerance Test in Patients With Type 2 Diabetes
Brief Title: The Effect of Exenatide Compared to Lantus Insulin on Vascular Function in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHS #05-45
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Results first posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: endothelial dysfunction; subclinical inflammation; flow mediated brachial artery dilation; pulse wave analysis; glucagon like polypeptide mimetics; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glargine insulin (Active Comparator): Glargine insulin 10-20 units once daily and subsequently adjusted per protocol to achieve fasting blood glucose of 100 mg/dl and avoid hypoglycemia.
  Interventions: Drug: Glargine Insulin
- Exenatide (Experimental): Exenatide 5ug twice daily for 4 weeks followed by 10 ug twice daily for 8 weeks.
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — Exenetide 5ug twice daily for 4 weeks, then 10ug twice daily for 8 weeks
  Other Names: Byetta
  Arms: Exenatide
Drug: Glargine Insulin — Glargine insulin 10-20 units once daily and subsequently adjusted per protocol to achieve a fasting glucose of 100mg/dl and avoid hypoglycemia.
  Other Names: Lantus insulin
  Arms: Glargine insulin

SUMMARY:
The main goals of the study are to evaluate the effect of Exenatide on endothelial-dependent vasodilation, as measured by flow mediated dilation (FMD), to evaluate the effect on endothelial-independent vasodilation, as measured by nitroglycerin (TNG) response, and to evaluate the effect on arterial stiffness, as measured by pulse wave analysis (PWA). We will also measure the effects on various markers of endothelial function, subclinical inflammation, fibrinolysis, and oxidative stress. The control group for the study will receive Lantus insulin, with a goal of similar glycemic control between the treatment and control groups.

Specific Aims

We will test the following hypotheses:

1. Treatment of patients with type 2 diabetes who are inadequately controlled by monotherapy with a Sulfonylurea (SU) or Metformin, or on combination therapy of a SU and Metformin with Exenatide (GLP-1 mimetic) will result in improved endothelial dependent vasodilation, as measured by FMD, as compared to the control group, who will be treated with Lantus insulin to achieve comparable HbA1c levels.
2. Treatment with Exenatide (GLP-1 mimetic) will result in improved arterial stiffness, as measured by AI by PWA, as compared to the control group, who will be treated with Lantus insulin to achieve comparable HbA1c levels.
3. Endothelial dependent vasodilation, as measured by FMD, and arterial stiffness, as measured by AI, measured in the postprandial state (following a standard test meal) will be improved following treatment with Exenatide as compared to treatment with once daily basal insulin (Lantus).
4. Treatment will result in no improvement in endothelial-independent vasodilation, as measured by a response to TNG, as compared to the control group, who will be treated with Lantus insulin to achieve comparable HbA1c levels.
5. Treatment with Exenatide, compared with treatment with Lantus, will result in a reduction in various plasma markers of inflammation (CRP, TNFA, IL6), endothelial activation (ICAM, VCAM, endothelin 1), fibrinolysis (PAI-1 protein, PAI-1 activity), and oxidative stress (FOX2).

DETAILED DESCRIPTION:
The trial is a randomized, controlled, comparator study. Subjects and investigators will not be blinded due to the nature of the treatment. After providing informed consent and meeting the inclusion and exclusion criteria, subjects will undergo baseline studies then be randomized to either treatment with Exenatide or Lantus insulin to achieve comparable improvement in glycemic control, as measured by HbA1c. A computer program (randomization.com) will be utilized to randomize 72 patients to receive either Exenatide or Lantus. The treatment group will receive twice daily injections of Exenatide, initially of 5ug BID, and increased to 10ug BID after 1 month. The control group will receive daily injections of Lantus insulin each evening, which will be titrated to achieve blood glucose targets based on self monitoring of blood glucose (SMBG), as outlined by the American Diabetes Association (ADA) (goal: fasting 90-130, peak postprandial less than180 mg/dl). The subjects on Lantus should achieve this goal by week 6 of the study, so that they have six weeks of maximal therapy. The control group will receive Lantus with the goal of similar glycemic control between the groups, with a goal of HbA1c reduction of 0.5-1.5% after 3 months. Based on recent data, it should be feasible to accomplish similar improvements in glycemia between the groups.

The trial will be preceded by a one-week screening and evaluation period, during which time the patient will be informed about the trial, and qualification will be determined based on the inclusion/exclusion criteria, as noted below. The patient will also be instructed in injection technique and SMBG techniques at the screening visit. Subjects will be asked to perform daily fasting blood glucose monitoring, and in addition on 2 days per week (1 weekday and 1 weekend day) to obtain 6 blood glucose measurements (fasting, 1-2hours post-breakfast, pre-lunch, 1-2 hours post-lunch, pre-dinner, and 1-2 hours post-dinner). Baseline studies will then be performed at week 0, including fasting laboratory studies, FMD, PWA, and Meal Challenge Test. The subject will then be randomized to receive treatment with either Lantus or Exenatide for 12 weeks duration. Repeat studies will then be performed at 12 weeks, including repeat of the baseline laboratory studies, FMD, PWA, and Meal Challenge test.

Schedule/Flow Chart

Visit 1 (week -1): Potential participants will be informed regarding the trial, records will be reviewed, and inclusion/exclusion criteria will be evaluated. Informed consent will be administered, and a history and physical will be performed. They will have baseline labs drawn, including HbA1c, glucose, lipids, CBC, chemistry, renal function, liver function, and urinalysis. If they are female and of reproductive age, they will also have a urine HCG performed. Subjects will be fasting for this visit.

Visit 2 (week 0): Participants will come in fasting. Interval medical history and medications will be reviewed. Vital signs will be obtained. PWA and FMD will be performed. The patient will then have fasting labs drawn which will include glucose, insulin, c-peptide, lipids, free fatty acids (FFA), CRP, TNFA, IL-6, ICAM, VCAM, endothelin 1, PAI-1 protein, PAI-1 activity, and FOX2. The patient will then have a mixed meal (time 0), and labs will again be drawn at 15, 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes, and 240 minutes after the meal challenge measuring glucose, insulin, c-peptide, lipids, and FFA. At time 120 minutes, FWA and FMD will be performed again along with blood samples for CRP, TNFA, IL-6, ICAM, VCAM, endothelin 1, PAI-1 protein, PAI-1 activity, and FOX2. At 240 minutes, PWA, FMD, and TNG will be performed.

After completion of these tests, the patients will be randomized and start treatment with either Exenatide 5ug BID or nightly Lantus beginning the following day. Lantus dose will be based on clinical assessment, but starting doses will likely be between 10 and 20 units. Patients will be instructed in SMBG techniques, as well as injection techniques for either Byetta (Exenatide) or Lantus.

Week 1: Telephone contact. Review side effects and blood glucoses (BGs), adjust Lantus if needed, and adjust oral hypoglycemic agents (OHA) in Exenatide treated group if clinically indicated.

Week 2: Telephone contact. Review side effects and BGs, adjust Lantus if needed, and adjust OHA in Exenatide treated group if clinically indicated.

Visit 3 (week 4): Patients will come in. Those in the Exenatide group will have the dose increased to 10ug sq BID. The patients in the Lantus group will have their fasting BGs reviewed and their dose adjusted. Side effects will be reviewed with all subjects. Subjects in the Exenatide treated group will have their OHA adjusted if clinically indicated.

Week 6: Telephone contact. Review BGs and side effects, and adjust Lantus if needed. Lantus dose should be at/close to maximal dose to achieve target fasting blood glucose goal. Subjects in the Exenatide treated group will have their OHA adjusted if clinically indicated.

Week 8: Telephone contact. Review side effects and BGs, adjust Lantus if needed, and adjust OHA in Exenatide treated group if clinically indicated.

Week 10: Telephone contact. Review side effects and BGs, adjust Lantus if needed, and adjust OHA in Exenatide treated group if clinically indicated. At this time, we will discuss with the subjects if they are interested in continuing their study medication upon completion of the study. We will advise them to call their diabetes provider to then arrange for a prescription that will start upon study completion. We will advise them at the beginning of the study to set up a follow up appointment with their provider around the time of study completion. We will speak with their diabetes provider if the subject wishes us to do so.

Visit 4 (week 12): Participants will come in fasting. If they are in the Exenatide group, we will ask them not to take their morning dose at home, but to bring it in with them so that it can be administered within 60 minutes of the meal tolerance test. Subjects will also be asked to return any unused study drug at this final visit. Interval medical history and medications will be reviewed. Vital signs will be obtained. PWA and FMD will be performed. The patient will then have fasting labs drawn which will include CBC, Chem 20, HbA1C, urinalysis, microalbumin, LFTs, glucose, insulin, c-peptide, lipids, FFA, CRP, TNFA, IL-6, ICAM, VCAM, endothelin 1, PAI-1 protein, PAI-1 activity, and FOX2. The subjects randomized to Exenatide will then take their morning dose, and all subjects will then have a mixed meal (time 0), and labs will again be drawn at 15, 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes, and 240 minutes after the meal challenge measuring glucose, insulin, c-peptide, lipids, and FFA. At time 120 minutes, PWA and FMD will be performed again along with labs for CRP, TNFA, IL-6, ICAM, VCAM, endothelin 1, PAI-1 protein, PAI-1 activity, and FOX2. At 240 minutes, PWA, FMD, and TNG will be performed.

Methods The Mixed Meal will consist of standard liquid meal, Boost, which is composed of 61.5g of carbohydrate, 15g of protein, and 6g of fat, in 360ml, with 360 calories. The subjects will come in fasting. Starting at time 0, the Boost will be consumed over a five minute time period. The studies will then be performed on visits 2 and 4.

Brachial artery flow mediated dilatation (FMD) evaluates endothelium-dependent reactivity in the macrocirculation. This is carried out in temperature-controlled room (24-26 degrees C) with a 30 minute acclimatization period. FMD of the brachial artery is measured at rest and during reactive hyperemia using a high-resolution 10.0 MHz linear array transducer and an HDI Ultramark 9 system. Reactive hyperemia is produced by inflating a pneumatic tourniquet distally to the brachial artery to 50 mmHg above the systolic BP for 5 minutes, then deflating it. Brachial artery diameter is measured before inflation of the cuff and 1-2 minutes after cuff deflation and expressed as the percentage change.

Trinitroglycerin-induced vasodilation evaluates endothelium independent vasodilation. The brachial artery will be scanned before and 5 minutes after sublingual administration of 400 ug of trinitroglycerin. This will be performed only at 240 minutes, fifteen minutes after completion of the FMD study to allow for the brachial artery to return to baseline.

Pulse wave analysis(PWA) is another method to evaluate the function of the vasculature. The shape of the arterial pressure waveform provides a measure of systemic arterial stiffness. All measurements will be made in the right arm using the Sphygmocore Px (Atcor Medical Blood Pressure Analysis System, Australia) in a temperature-controlled room. With the wrist slightly extended and supported on a pillow, the radial artery of the right arm is flattened with a high fidelity micro manometer using gentle pressure. 20 sequential waveforms are acquired and the system software generates an average peripheral and corresponding central waveform, which is then subjected to further analysis of augmentation. Two pressure peaks characterize the systolic part of the central waveform. The first peak results from LV ejection, and the second results from the wave reflection. The difference between peaks represents the degree to which central arterial pressure is augmented by wave reflection. AP is the absolute increase in pressure from the reflected wave and AI is a measure of the contribution that the wave reflection makes to the arterial pressure waveform, and is expressed as a percentage of pulse pressure. The amplitude and timing of the reflected wave ultimately depends on the stiffness of the small vessels and large arteries, and thus is a measure of systemic arterial stiffness.

We will enroll 72 subjects to obtain 60 subjects who will complete the study. The subjects will have Type 2 diabetes and will be randomized to one of two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75
* Type 2 Diabetes (diagnosed at least 3 months prior to study)
* HbA1c: above 7.0 and less than or equal to 10.0
* At least one HbA1c over preceding 3-6 months, and HbA1c at screening, with less than 1% difference between lowest and highest values
* Stable doses of antidiabetic medications (SU and/or Metformin) for 3 months
* reproductive age females must have negative urine HCG at screening, and be using appropriate contraception during the study or be surgically sterile
* postmenopausal woman
* stable weight for 3 months prior to study (+/- 2kg)
* willingness to participate in the study

Exclusion Criteria:

* Type 1 diabetes
* Type 2 diabetes less than 3 months in duration
* HbA1c less than 7.0 or greater than 10
* age less than 18 or greater than 75
* pregnant or planning to become pregnant during study period
* current insulin therapy or insulin within 6 months prior to study
* current use of Thiazolidinedione or within 6 months prior to study
* current use of Nateglinide or Repaglinide
* current use of an Alpha-glucosidase Inhibitor
* current weight loss program
* active smoker, or quit smoking within preceding 6 months
* creatinine greater than 2.0 mg/dL
* total cholesterol greater than 300 mg/dL
* triglycerides greater than 600 mg/dL
* blood pressure greater than 160/105 mmHg
* ALT/AST greater than twice the upper limit of normal
* any other medical condition that may interfere with trial participation or trial results
* if on Statin: Statin therapy for less than 3 months or dose change within preceding 3 months
* if on ACE Inhibitor: ACE Inhibitor therapy for less than 3 months or dose change within preceding 3 months
* current use of any medication that is known to alter gastric motility

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward S. Horton, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Joslin Diabetes Center Clinic, Boston, MA, from July 2006-0ctober 2009. Subjects had Type 2 diabetes, treated with either Metformin, SU, Metformin/SU, TZD, or Metformin/TZD, on stable therapy and weight for 3 months.
  The healthy controls in the Extension Study, were recruited from the Joslin Diabetes Center.
Pre-assignment Details: Baseline fasting studies on all subjects included anthropometrics, blood pressure, HbA1c, glucose, insulin, c-peptide, lipids, free fatty acids (FFA), hsCRP, TNFa, IL-6, siCAM, sVCAM, PAI-1 antigen, and oxidized LDL. PWA and FMD were measured fasting and after a standardized meal with repeat PWA and FMD at 2 and 4 hours, and TNG at 4 hours.
Period: Overall Study
Arm/Group | Glargine Insulin | Exenatide
Started | 26 | 27
Completed | 26 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glargine Insulin | Exenatide | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 27 | 53
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (8.5) | 58.4 (11.6) | 59.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 16 | 15 | 31
Region of Enrollment [Number; unit: participants]
  United States | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint Was the Change in FMD at the End of the Study Compared to Baseline Measurements in Subjects Treated With Exenatide Compared to Subjects Treated With Lantus.
Description: Flow mediated dilation (FMD) of the brachial artery was measured at rest and during reactive hyperemia using a high-resolution 10.0 MHz linear array transducer and an HOI Ultramark 9 system. Reactive hyperemia was produced by inflating a pneumatic tourniquet on the forearm distal to the brachial artery to 50 mmHg above the systolic BP for 5 minutes, then deflating it . Brachial artery diameter was measured before inflation of the cuff and 1-2 minutes after cuff deflation and expressed as the percentage change. This protocol is described in detail elsewhere. This was performed fasting, 2, and 4 hours after the meal challenge at baseline and 3 months.
Time Frame: Baseline and End of Study
Measure: Mean (Standard Deviation); unit: Percentage dilation
Arm/Group | Glargine Insulin | Exenatide
Number analyzed (Participants) | 26 | 27
Percentage dilation | 5.0 (2.3) | 4.7 (2.4)

2. Secondary Outcome: First Will be the Changes in TNG Stimulated Arterial Dilation (Endothelial-independent) in Subjects Treated With Exenatide Compared With Subjects Treated With Lantus at the End of the Study Compared to Baseline Measurements
Description: Trinitroglycerin (TNG) response evaluates endothelium independent vasodilation. The brachial artery was scanned before and 5 minutes after sublingual administration of 400 ug of trinitroglycerin. This was performed only at 4 hours following the test meal and fifteen minutes after completion of the FMD study to allow for the brachial artery to return to baseline. This was performed at both the baseline and 3 month visits.
Time Frame: Baseline and end of study
Measure: Mean (Standard Deviation); unit: Percentage dilation
Arm/Group | Glargine Insulin | Exenatide
Number analyzed (Participants) | 26 | 27
Percentage dilation | 10.7 (5.3) | 11.3 (4.5)

3. Secondary Outcome: Second Will be the Change in Arterial Stiffness, as Measured by PWA, in Subjects Treated With Exenatide Compared With Subjects Treated With Lantus at the End of the Study Compared to Baseline Measurements.
Time Frame: Baseline and end of study
Reporting Status: Not Posted

4. Secondary Outcome: Third Will be the Changes in Markers of Endothelial Function, Inflammation, Fibrinolysis, and Oxidative Stress in Subjects Treated With Exenatide Compared With Subjects Treated With Lantus at the End of the Study Compared to Baseline
Time Frame: Baseline and end of study
Reporting Status: Not Posted

5. Secondary Outcome: Fourth Will be Changes in Insulin, Glucose, C-peptide, Lipids, and FFA Responses Following the MTT in Subjects Treated With Exenatide Compared With Subjects Treated With Lantus at the End of the Study Compared to Baseline Measurement
Time Frame: Baseline and end of study
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 years and 3 months
Description: No adverse events reported
Arm/Group | Glargine Insulin | Exenatide
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 0/26 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No